CLINICAL TRIAL: NCT02589847
Title: An Open-label Efficacy and Safety Assessment of Rebiotix RBX2660 (Microbiota Suspension) for the Treatment of Recurrent Clostridium Difficile Infection
Brief Title: Microbiota Restoration Therapy for Recurrent Clostridium Difficile Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rebiotix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-01
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Results first posted 2020-05-11 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-02

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; C diff; CDI; CDAD; Fecal transplant; Fecal Microbiota transplant; diarrhea; FMT; microbiota restoration therapy; microbiota suspension; fecal bacteriotherapy; C diff diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RBX2660 Open-label (Experimental): RBX2660 (microbiota suspension)
  Interventions: Biological: RBX2660
- Historical control antibiotics (Other): Retrospective Historical Control with standard of care
  Interventions: Drug: Standard of Care Antibiotics

INTERVENTIONS:
Biological: RBX2660 — suspension of intestinal microbes
  Arms: RBX2660 Open-label
Drug: Standard of Care Antibiotics — Standard of Care Antibiotics
  Other Names: Antibiotics
  Arms: Historical control antibiotics

SUMMARY:
This study will evaluate efficacy and safety information about RBX2660 for the treatment of recurrent Clostridium difficile infection (CDI), and will compare the efficacy of one treatment with RBX2660 versus antibiotic-treated historical controls. Enrolled subjects will receive one treatment consisting of two doses of RBX2660 (microbiota suspension).

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label study assessing the efficacy and safety of RBX2660 as an adjunct to antibiotics for the treatment of recurrent CDI. Efficacy of RBX2660, measured by the recurrence-free rate of CDI diarrhea without the need for retreatment with C. difficile anti-infective therapy or fecal transplant through 56 days after completion of study treatment with RBX2660, will be evaluated by comparing the recurrence-free rate observed in the study population to the recurrence-free rate identified from antibiotic-treated historical controls.

Patients who have had either a) at least two recurrences after a primary episode (i.e., at least three episodes) and have completed at least two rounds of standard-of-care oral antibiotics or b) have had at least two episodes of severe CDI resulting in hospitalization may be eligible to participate in the study. Study visits are 1- and 8-weeks after treatment with additional follow-up assessments at 3,6,12, and 24 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old.
* Medical record documentation of recurrent CDI including a positive C. difficile test within 60 days prior to enrollment and either: a) at least two recurrences after a primary episode and has completed at least two rounds of standard-of-care oral antibiotic therapy or b) has had at least two episodes of severe CDI resulting in hospitalization.
* Documented history that the subject's recurrent CDI is controlled while on antibiotics even if the subject is not currently on antibiotics.
* A positive stool test for the presence of C. difficile within 60 days prior to enrollment

Exclusion Criteria:

* A known history of continued CDI diarrhea despite being on a course of antibiotics prescribed for CDI treatment.
* Requires continuous antibiotic therapy for a condition other than CDI.
* Previous successful (resolution of CDI diarrhea) fecal transplant for recurrent CDI < 6 months prior to study enrollment.
* Previous unsuccessful (recurrent CDI diarrhea was unresolved) fecal transplant.
* Previous treatment with RBX2660.
* Diagnosis of inflammatory bowel disease (IBD), e.g., ulcerative colitis, Crohn's disease, or microscopic colitis.
* Diagnosis of irritable bowel syndrome (IBS) as determined by Rome III criteria.
* History of chronic diarrhea.
* History of celiac disease.
* Disease symptoms caused by a confirmed intestinal pathogen other than C. difficile.
* Colostomy.
* Planned surgery requiring perioperative antibiotics within 3 months of study enrollment.
* Life expectancy of < 12 months.
* Compromised immune system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Ray, MD, Study Chair — Ochsner Health System
Locations (30):
- United States (28):
  - Phoenix, Arizona
  - North Little Rock, Arkansas
  - Sacramento, California
  - Bay Pines, Florida
  - Coral Springs, Florida
  - Gainesville, Florida
  - Miami, Florida
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Maywood, Illinois
  - Indianapolis, Indiana
  - Lafayette, Indiana
  - Lexington, Kentucky
  - Detroit, Michigan
  - Rochester, Minnesota
  - Saint Paul, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Flushing, New York
  - Rochester, New York
  - Syracuse, New York
  - The Bronx, New York
  - Fargo, North Dakota
  - Lima, Ohio
  - Jackson, Tennessee
  - Houston, Texas
  - Springfield, Virginia
  - Virginia Beach, Virginia
- Canada (2):
  - Vancouver, British Columbia
  - Hamilton, Ontario

REFERENCES:
- [Derived] Lee C, Feuerstadt P, Louie T, Bancke L, Guthmueller B, Harvey A, Hoeyer F, Orenstein R, Dubberke ER, Khanna S. Integrated analysis of the safety of fecal microbiota, live-jslm in adults with recurrent Clostridioides difficile infection from five prospective clinical trials: an update. Therap Adv Gastroenterol. 2025 Nov 12;18:17562848251395566. doi: 10.1177/17562848251395566. eCollection 2025. PMID 41245385
- [Derived] Reveles KR, Gonzales-Luna AJ, Golan Y, Alonso CD, Guthmueller B, Tan X, Bidell MR, Pokhilko V, Crawford CV, Skinner AM. Efficacy of Fecal Microbiota, Live-jslm (REBYOTA(R)), Among Patients Exposed to Non-Clostridioides difficile Infection Antibiotics: Post Hoc Subgroup Analysis of a Phase 2 Open-Label Study. Open Forum Infect Dis. 2024 Jun 17;11(7):ofae341. doi: 10.1093/ofid/ofae341. eCollection 2024 Jul. PMID 39006315
- [Derived] Orenstein R, Dubberke ER, Khanna S, Lee CH, Yoho D, Johnson S, Hecht G, DuPont HL, Gerding DN, Blount KF, Mische S, Harvey A. Durable reduction of Clostridioides difficile infection recurrence and microbiome restoration after treatment with RBX2660: results from an open-label phase 2 clinical trial. BMC Infect Dis. 2022 Mar 12;22(1):245. doi: 10.1186/s12879-022-07256-y. PMID 35279084

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RBX2660 Open-label | Historical Control Antibiotics
Started | 162 | 110
Safety Population | 149 | 0
Full Analysis Set (FAS) | 149 | 104
Evaluable | 142 | 75
Completed | 107 | 39
Not Completed | 55 | 71

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | RBX2660 Open-label | Historical Control Antibiotics | Total
Number analyzed (Participants) | 149 | 104 | 253
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 40 | 102
  >=65 years | 87 | 64 | 151
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 71 | 166
  Male | 54 | 33 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 142 | 44 | 186
  Unknown or Not Reported | 3 | 55 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 136 | 40 | 176
  More than one race | 0 | 16 | 16
  Unknown or Not Reported | 3 | 45 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were CDI-diarrhea Free Through 8 Weeks
Description: Participants were evaluated 8 weeks after study treatment to assess efficacy of RBX2660. Efficacy was assessed as the absence of CDI diarrhea without the need for retreatment with C. difficile anti-infective therapy or fecal transplant through 56 days after completion of study treatment.
Time Frame: 8 weeks after treatment
Population: Evaluable Population - All participants evaluable for a treatment outcome through 56 days after completion of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | RBX2660 Open-label | Historical Control Antibiotics
Number analyzed (Participants) | 142 | 75
Participants
  Treatment Success | 112 | 23
  Treatment Failure | 30 | 52

2. Secondary Outcome: Quality of Life (SF-36)
Description: The Short Form - 36 quality of life questionnaire (SF-36) is a tool used to identify changes to quality of life following study treatment. It consists of a series of 36 questions relating to Mental and Physical health, summarized by a Physical Component Score (PCS) and Mental Component Score (MCS), respectively. Several sub-scales exist for each of the larger components; PCS includes PF, RP, BP, and GH while, MCS includes VT, SF, RE, and MH [All abbreviations are defined in table]. All Sub-Scale and Component Scores were calculated using Quality Metric Health Outcomes Scoring Software v4.5. The range of all scores is normalized from 0 (worst) to 100 (best). The data is presented for mean scores at baseline and 8-weeks post-treatment.
Time Frame: Baseline
Population: Safety Population - The SP includes all participants who were enrolled and received at least dose of RBX2660.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RBX2660 Open-label
Number analyzed (Participants) | 149
score on a scale
  Physical Component Summary (PCS): number analyzed (Participants) | 137
  Physical Component Summary (PCS) | 40.3 (9.3)
  Physical Functioning (PF): number analyzed (Participants) | 143
  Physical Functioning (PF) | 39.8 (11.8)
  Role Limitations Due to Physical Health (RP): number analyzed (Participants) | 147
  Role Limitations Due to Physical Health (RP) | 38.0 (11.3)
  Bodily Pain (BP): number analyzed (Participants) | 147
  Bodily Pain (BP) | 44.5 (11.5)
  General Health Perceptions (GH): number analyzed (Participants) | 147
  General Health Perceptions (GH) | 44.6 (10.7)
  Mental Component Summary (MCS): number analyzed (Participants) | 137
  Mental Component Summary (MCS) | 45.5 (12.3)
  Vitality (VT): number analyzed (Participants) | 145
  Vitality (VT) | 41.9 (11.5)
  Social Functioning (SF): number analyzed (Participants) | 145
  Social Functioning (SF) | 40.1 (12.2)
  Role Limitations Due to Emotional Problems (RE): number analyzed (Participants) | 144
  Role Limitations Due to Emotional Problems (RE) | 43.6 (12.2)
  Mental Health (MH): number analyzed (Participants) | 144
  Mental Health (MH) | 46.3 (11.7)

3. Secondary Outcome: Quality of Life (SF-36)
Description: as for outcome 2
Time Frame: 8-Weeks
Population: Safety Population - The SP includes all participants who were enrolled and received at least dose of RBX2660.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RBX2660 Open-label
Number analyzed (Participants) | 149
score on a scale
  Physical Component Summary (PCS): number analyzed (Participants) | 106
  Physical Component Summary (PCS) | 44.3 (11.1)
  Physical Functioning (PF): number analyzed (Participants) | 113
  Physical Functioning (PF) | 42.2 (12.6)
  Role Limitations Due to Physical Health (RP): number analyzed (Participants) | 114
  Role Limitations Due to Physical Health (RP) | 43.8 (10.7)
  Bodily Pain (BP): number analyzed (Participants) | 112
  Bodily Pain (BP) | 48.6 (11.8)
  General Health Perceptions (GH): number analyzed (Participants) | 111
  General Health Perceptions (GH) | 48.0 (10.0)
  Mental Component Summary (MCS): number analyzed (Participants) | 106
  Mental Component Summary (MCS) | 50.9 (10.4)
  Vitality (VT): number analyzed (Participants) | 113
  Vitality (VT) | 49.0 (10.5)
  Social Functioning (SF): number analyzed (Participants) | 111
  Social Functioning (SF) | 47.2 (11.3)
  Role Limitations Due to Emotional Problems (RE): number analyzed (Participants) | 114
  Role Limitations Due to Emotional Problems (RE) | 46.9 (11.8)
  Mental Health (MH): number analyzed (Participants) | 111
  Mental Health (MH) | 51.0 (10.6)

4. Secondary Outcome: Number of Participants With Major Complications of rCDI From Baseline Through 24 Months
Description: Major complications of rCDI, defined as death, septic shock, toxic megacolon, colonic perforation, emergency colectomy, or ICU admission) were collected and reported as a safety-related endpoint.
Time Frame: 24 months
Population: Full Analysis Set- Defined as participants who received at least one dose of RBX2660 or was in the Historical Control Arm
Measure: Count of Participants; unit: Participants
Arm/Group | RBX2660 Open-label | Historical Control Antibiotics
Number analyzed (Participants) | 149 | 104
Participants
  At least one complication of rCDI | 3 | 2
  Death | 1 | 0
  Septic Shock | 2 | 1
  Toxic Megacolon | 0 | 0
  Colonic Perforations | 0 | 0
  Emergency Colectomy | 0 | 1
  ICU Admission | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from enrollment through 24 months after treatment for participants who received RBX2660. Historical Control subjects were followed for up to 6 months.
Description: Treatment emergent adverse events are presented, defined as adverse events that occurred after exposure to study drug.
  For participants that received RBX2660, at each contact point (in office visit or scheduled phone call) they were systematically asked about adverse events, as well as use of a subject diary for one week post the last study enema.
Arm/Group | RBX2660 Open-label | Historical Control Antibiotics
All-Cause Mortality (participants affected / at risk) | 15/149 | 5/104
Serious Adverse Events (participants affected / at risk) | 52/149 | 30/104
Other Adverse Events (participants affected / at risk) | 118/149 | 62/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RBX2660 Open-label (N=149) | Historical Control Antibiotics (N=104)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 5 (5) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 6 (11) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 2 (2)
Sepsis (Infections and infestations) | 8 (10) | 3 (3)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 3 (3) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 2 (2) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 3 (3) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydroureter (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 3 (4) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Hypertensive crisis (Vascular disorders) | 2 (3) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 3 (5)
Colitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Vital functions abnormal (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Dilatation ventricular (Cardiac disorders) | 1 (1) | 0 (0)
Cogan's syndrome (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 4 (4) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dialysis related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0)
Staphylococcus test positive (Investigations) | 1 (1) | 0 (0)
Venous pressure jugular increased (Investigations) | 1 (1) | 0 (0)
Inflammatory marker increased (Investigations) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium tremens (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Immobile (Social circumstances) | 1 (1) | 0 (0)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0)
Diffuse vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RBX2660 Open-label (N=149) | Historical Control Antibiotics (N=104)
Diarrhoea (Gastrointestinal disorders) | 42 (69) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 18 (30) | 1 (1)
Flatulence (Gastrointestinal disorders) | 8 (9) | 1 (1)
Constipation (Gastrointestinal disorders) | 17 (21) | 4 (9)
Abdominal distension (Gastrointestinal disorders) | 9 (11) | 1 (2)
Nausea (Gastrointestinal disorders) | 10 (15) | 2 (2)
Urinary tract infection (Infections and infestations) | 17 (20) | 17 (22)
Headache (Nervous system disorders) | 9 (9) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (10)
Dizziness (Nervous system disorders) | 2 (2) | 6 (7)
Fatigue (General disorders) | 3 (4) | 9 (9)
Asthenia (General disorders) | 4 (4) | 7 (8)
Oedema peripheral (General disorders) | 2 (3) | 6 (11)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT02589847/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT02589847/SAP_001.pdf